CLINICAL TRIAL: NCT04200833
Title: Golimumab in Juvenile Idiopathic Arthritis-associated Uveitis Failing Adalimumab
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 31-301ex18/19
Record Dates: First submitted 2019-08-06; First posted 2019-12-16 (Actual); Results first posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: JIA Associated Uveitis
Keywords: Biological; Uveitis; adalimumab; golimumab
MeSH Terms: conditions — Uveitis | interventions — golimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group 1: All JIA patients that were switched from adalimumab to golimumab because of Treatment failure of their JIA associated uveitis at the Medical University of Graz Austria from 2010 to 2019
  Interventions: Drug: Golimumab

INTERVENTIONS:
Drug: Golimumab — subcutaneous injection

SUMMARY:
To asses the use of golimumab, a fully humanized anti-TNF Alpha monoclonal antibody, in juvenile idiopathic Arthritis-associated uveitis refractory to adalimumab.

DETAILED DESCRIPTION:
Background:

Uveitis is a potentially blinding complication of juvenile idiopathic arthritis (JIA). Treatment remains a substantial challenge, even though the use of tumor necrosis factor (TNF)-α-antagonists has improved visual outcomes substantially. Among these agents, adalimumab has been recently approved for the treatment of non-infectious uveitis and is thus the first biologic disease-modifying anti-rheumatic drug (bDMARD) approved for JIA-associated uveitis. However, some patients do not respond sufficiently or lose response over time. In these cases switching to another biologic DMARD is recommended. Recently golimumab, a fully humanized anti-TNF-α monoclonal antibody, demonstrated efficacy in a small case series, leading to uveitis inactivity in 4 of 7 patients Golimumab is approved for the treatment of polyarticular JIA.

Hypothesis:

Patients with JIA-associated uveitis failing treatment with adalimumab benefit from the treatment with golimumab.

Methods:

Study design and patient recruitment (retrospectively)

Retrospective single-center study in patients with JIA-associated active uveitis at the Medical University of Graz/Austria, in whom golimumab was started after failure of standard conventional immunosuppressive drugs and adalimumab. All patients that have started golimumab from March 2010 are included in the study. Uveitis is defined and anatomically classified according to the recommendations of the Standardization of Uveitis Nomenclature (SUN) Working Group. Primary failure to adalimumab was diagnosed in patients without change in the SUN score and an entry grade of 3 or higher or with worsening activity, defined as either a two-grade increase in inflammation or an increase to grade 4. With bilateral disease, the eye with the higher grade of uveitis was analysed. Relapse of uveitis was defined as active inflammation after an inactivity for at least 3 months. Loss of response was defined as failure to improve under continued treatment with adalimumab despite intermitting intensifying concomitant therapy, such as local or systemic steroids.

Golimumab treatment was administered in the standard dose of 50 mg sc every 4 weeks in patients with a weight of at least 40 kg. Previous therapy with a conventional DMARD such as methotrexate (MTX) was continued, if tolerated.

The outcome measures of uveitis include the reduction in grade of intraocular inflammation, the best-corrected visual acuity, eye soreness, redness of eyes, light sensitivity and the steroid sparing potential. Response to treatment is classified as complete, partial or no response. Complete response constitute achieving inactive uveitis, defined as <0.5 cell per field in the anterior chamber or posterior segment (grade 0) and absence of vitreous haze and macular edema. Partial response is diagnosed in patients with improved uveitis, defined as decrease of one grade in the level of inflammation, without a decrease to grade 0 in the anterior chamber (AC) and posterior segment. Primary failure, relapse and loss of response to golimumab is defined in the same way as for adalimumab.

Patients receiving Golimumab were evaluated clinically and immunologically at regular intervals. At each visit the laboratory analysis included complete blood cell counts, levels of creatinine, hepatobiliary-injury biomarkers, and C-reactive protein. Side effects were assessed by patient's reported history.

Statistical analysis Continuous variables will be analyzed by Student's t-test or Mann-Whitney U test. Correlations will be analyzed by Spearman's rank correlation test. Binary variables were analyzed using Fisher's exact test. Statistical significance was defined as p<0.05. All statistical analyses were performed using GraphPad Prism V.6.0 (GraphPad, San Diego, CA).

ELIGIBILITY:
Inclusion Criteria:

* JIA associated Uveitis
* Treatment failure with adalimumab

Exclusion Criteria:

* Uveitis due to other causes
* Adalimumab Initiation because of non ocular reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: JIA patients at a tertiary referal Center in Graz /Austria. University setting.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reported as Complete Responders to Golimumab
Description: Response was classified as complete, partial, or none ("non-response", NR) at each timepoint separately." Complete response (CR) constituted achieving inactive uveitis, defined as 0+ cells in the AC (grade 0). Partial response (PR) was diagnosed in patients with improved uveitis, defined as a decrease in the level of inflammation, without achieving AC grade 0 status. Primary-NR was diagnosed in patients without change in SUN score and an entry grade of 3 or higher or in patients with worsening activity, defined as either a two-grade increase in inflammation or an increase in inflammation to grade 4. Relapse of uveitis was defined as active inflammation after at least 3 months of inactivity,
Time Frame: last follow up, up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1
Number analyzed (Participants) | 10
Participants | 8

2. Secondary Outcome: Best Corrected Visual Acuity (BCVA)
Description: best corrected visual acuity
Time Frame: up to 5 years
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Group 1
Number analyzed (Participants) | 10
LogMAR | 0.27 (0.33)

3. Secondary Outcome: Number of Patients With Ocular Discomfort
Description: eye soreness, photophobia
Time Frame: up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1
Number analyzed (Participants) | 10
Participants | 0

4. Secondary Outcome: Steroid Sparing Potential
Description: Reduction in systemic steroid dose at the 12 month follow-up compared to baseline
Time Frame: Baseline, 12 Months Follow-Up
Measure: Mean (Full Range); unit: mg/kg per day
Arm/Group | Group 1
Number analyzed (Participants) | 10
mg/kg per day | 0.19 [0 to 0.52]

ADVERSE EVENTS:
Time Frame: Up to 66 months
Arm/Group | Group 1
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT04200833/Prot_SAP_000.pdf